CLINICAL TRIAL: NCT06874894
Title: Thromboembolic and Bleeding Risk During Anticoagulant Treatment in Asian Patents With Atrial Fibrillation
Brief Title: Thromboembolic And Bleeding Risks During anticoaGulant trEatment in Asian paTients With Atrial Fibrillation (TARGET-AF)
Acronym: NOAC
Status: Enrolling by invitation | Type: Observational
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Collaborators: Chung-Ang University Gwangmyeong Hospital (Other); Samsung Medical Center (Other); Korea University Ansan Hospital (Other); Kosin University Gospel Hospital (Other); Keimyung University Dongsan Medical Center (Other); Yuhan Corporation (Industry)
Responsible Party: Principal Investigator, Ki-Woon Kang, Associate Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Other Study IDs: CAUH 1992-002-387
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Fibrillation, Atrial
Keywords: Atrial Fibrillation; Stroke; Bleeding
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial Fibrillation: Documented AF on 12-lead ECG, Holter monitoring, or single-lead ECG recordings and biomarkers using TEG®-6S with NOAC treatment

SUMMARY:
This study was design to investigate the efficacy and safety of NOAC therapy in Koreans

DETAILED DESCRIPTION:
East Asians have demonstrated a higher bleeding tendency compared to Western populations during an anticoagulation. Consequently, East Asians have been prescribed as a relatively weaker treatment regimens based on this evidence. Therefore, the TARGET-AF study aims to verify the efficacy and safety of NOAC therapy using biomarkers including TEG®-6S point-of-care device in Koreans

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented AF on 12-lead ECG, Holter monitoring, or single-lead ECG recordings are eligible for enrollment.
* Based on AF treatment Korean guideline 19, AF patients who require NOAC treatment or are currently on NOAC treatment (within the past 3 months)
* Adults aged 18 or above who have provided consent for clinical information

Exclusion Criteria:

* Patients with moderate or severe mitral stenosis or mechanical prosthetic valve

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AF patients with NOAC
Sampling Method: Non-Probability Sample
Enrollment: 1021 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Clinical ischemic and hemorrhagic events | 12 months
  The Rate of Ischemic stroke, systemic embolism, or myocardial infarction and ISTH (International Society on Thrombosis and Hemostasis) major/minor bleeding events

SECONDARY OUTCOMES:
Clinical other events | 12 months
  The rate of Major Adverse Cardiovascular Events: Myocardial infarction, ischemic stroke, systemic embolism, and cardiovascular death (including bleeding).

OTHER OUTCOMES:
COVID-19 infection | 12 months
  The rate of confirmation of COVID-19 infection and primary outcome

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
CAUH 1992-002-387
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Lee SH, Kim HK, Ahn JH, Kang MG, Kim KH, Bae JS, Cho SY, Koh JS, Park Y, Hwang SJ, Gorog DA, Tantry US, Bliden KP, Gurbel PA, Hwang JY, Jeong YH. Prognostic impact of hypercoagulability and impaired fibrinolysis in acute myocardial infarction. Eur Heart J. 2023 May 14;44(19):1718-1728. doi: 10.1093/eurheartj/ehad088. PMID 36857519